CLINICAL TRIAL: NCT05399719
Title: Targeting Fusion Machinery Between Macrophages and Cancer Cells to Ameliorate Cancer Desmoplasia
Brief Title: Cancer Fusion Hybrids and Desmoplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: 202201057RINA
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2023-06

CONDITIONS: Fusion Protein Expression; Bone Marrow Cells
Keywords: fusion hybrids, macrophages, cancer cells

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — paraffin section of tumor tissues, peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tumor tissue from BMT recipients: tumor tissue sections from patients received allogeneic bone marrow transplantation before
- Peripheral blood from healthy volunteer: peripheral blood from peripheral blood stem cell donors or healthy control

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
Clinical and preclinical evidence reveal that cancer cells may fuse with hematopoietic cells to obtain properties including migration, proliferation and drug resistance. The investigators hypothesize that cancer cell-macrophage fusion hybrids may lead to pancreatic cancer desmoplasia and progression.

Murine tumor models using cre-loxP or gender-mismatched xenografts as well as pdx-cre-KrasLSL-G12D mice after bone marrow transplantation from reporter ROSA mice were established. Fusion hybrids and macrophage markers were detected using immunofluorescence staining and flowcytometry.

In vitro co-culture using cre-loxP or dual fluorescence methods of pancreatic cancer cells with macrophages was used to evaluate the frequency of fusion phenomenon. The proliferative, migratory and resistant phenotypes of purified fusion hybrids were measured. Differentially expressed genes between fusion hybrids and non-fused cancer cells were compared by Affymetrix microarray analysis.

The investigators are going to collect tumor tissues from cancer patients who received allographic bone marrow transplantation before. We will evaluate Y chromosome or short tandem repeats to identify donor- derived genes in cancer cells and demonstrate the clinical evidence of fusion between cancer cells and macrophages. The tumor tissues will be collected from the Pathology Department. Ten slides of 4-8um will be collected from twenty patients enrolled according to the inclusion criteria.

The investigator will collect peripheral mononuclear cells from healthy volunteer ( eg. Donors for bone marrow transplantation) or hyperemia patients. The mononuclear cells will be induced to differentiate into macrophages and will be co-cultured with cancer cells in order to purify fusion hybrids. The fusion hybrids between cancer cells and macrophages will be evaluated for biologic characters including proliferation, radio-sensitivity, migration etc. The investigators planned to collect blood samples from Department of Laboratory Medicine, Blood bank. Thirty subjects of healthy volunteer or hyperemia patients will be enrolled. Ten to 20ml peripheral blood will be collected from each subjects for one time.

DETAILED DESCRIPTION:
Desmoplasia has been shown to exert mechanical forces and create a biochemical intra-tumoral immunity and influence the development and progression of a malignancy. Recent reports suggest a significant negative correlation between cancer patient survival and extracellular matrix deposition in primary tumors; and concomitant stromal targeting may enhance therapeutic outcomes in cancer patients.

In defining the source of the dense stroma, it is generally believed that over-activated CAFs could produce extracellular matrix (ECM) proteins, the major component of the dense stroma. Anti-fibrosis drugs including those depleting CAFs or collagen, sonic hedgehog inhibitor, antibodies against LOX/LOX2, were under clinical trials. However, CAF-depleted tumors displayed a more aggressive phenotype and alteration in regulatory T cells, raising the possibility that CAF-targeting strategies may have both beneficial and detrimental effects.

Considering the functional significance of macrophages in inflammation, desmoplasia, cancer initiation and progression, mounting studies had conducted to evaluate the efficiency of anti-macrophage as a novel strategy against cancer. Accordingly, the anti-macrophage strategies include the inhibition of the monocytes recruitment as well as transformation, and the ablation the macrophages directly. Given the multifaceted roles of maintaining homeostasis, the systemic depletion of macrophages may lead to increased infections or impaired ability of tissue-resident cells to carry out their normal function. Thus, the identification of tumor associated macrophage (TAM)-specific markers will enable the development of more sophisticated therapies that can be targeted specifically to tumors without affecting the function of other tissue-resident immune cells.

Recent studies had identified numerous factors such as platelet-derived growth factor (PDGF) and transforming growth factor b1 (TGFb1) released by TAMs, especially bone marrow (BM)-derived ones, involving in the process of activating CAFs. In addition, there were TAMs-derived pro-fibrotic factors, such as connective tissue growth factor (CTGF), chemokine ligand 17 (CCL17), CCL22 and reactive oxygen species (ROS). Similar observation was found in TAMs-derived matrix metallopeptidase 9 (MMP9) which involved in the stroma turnover by degrading the ECM proteins. However, rare study investigates the role of fusion between macrophages and cancer cells in desmoplasia and tumor progression as well as the strategy targeting fusion machinery of macrophages with cancer cells.

Several lines of evidence support that cell fusion between cancer cells and leukocytes, majorly macrophages, is one of the explanations for tumor resistance and progression. Recent genotyping of a metastatic melanoma to the brain that arose following allogeneic BM transplantation supports, first time clinically, fusion between a BM derived cell and a tumor cell playing a role in the origin of metastasis. Fusion hybrids enumerated in peripheral blood of pancreatic cancer patients were reported to correlate with disease stage and predict overall survival. Furthermore, general inflammatory responses were demonstrated to increase the number of fusion events. While the fusion events were demonstrated in animal and human, and were correlated with cancer resistance and metastasis, little is known regarding key questions such as the mechanisms through which macrophage-cancer cell fusion and subsequent genomic hybridization occurs in vivo; potential survival advantages of hybrids; reprogramming of fibrotic and immunologic tumor microenvironment by hybrids; and the development of novel strategies to target fusion machinery.

The majority of macrophages, including tissue macrophages in normal tissue and TAMs, are derived from bone marrow (BM). The investigators' preliminary study, using irradiated murine intestine model, suggested parallel between the development of cell fusion between BM-derived monocytes and intestine stromal cells with radiation-induced fibrosis. Using cre-loxP system and gender mismatched BM transplantation, we demonstrated that BM-derived CD11b(+) myelo-monocytic cells/macrophages were the major fusion partner to damaged intestine stromal cells after radiation. The fusion events in irradiated intestine stroma correlated with chronic intestine fibrosis with enhanced TGFb transcripts and collagen deposition. With macrophage deletion by liposomal clodronate or conditional CD11b knock-out, we can ameliorate radiation induced chronic intestine fibrosis.

The main property of cancer cells that makes them malignant is the ability to produce diverse progeny. Fusion between cancer cells and TAMs can be an engine of genomic and epigenetic variability that has a potential to make cells with new properties at a rate exceeding that achievable by random mutation. Previous reports revealed cell fusion contribute to drug resistance and can promote the ability of cancer cells to metastasize.

Fibrosis and inflammation are hallmarks of tumor desmoplasia. TAMs, majorly derived from bone marrow,5 act as an essential connecting moiety between inflammation and cancer via secretion of pro-inflammatory cytokines/chemokines. The M2 polarized macrophages, which constitute majority of the macrophages in tumor microenvironment, secrete IL10 and other cytokines that mediate T helper 2 (Th-2) responses and are responsible for malignant tumor transformation and inhibit antitumor immune response mediated by T cells. TAMs were reported to play a phenomenal role in enhancing mesenchymal phenotype of cancer cells via TGFb. The lipopolysaccharide (LPS) receptor toll-like receptor 4 (TLR4) on the surface of TAMs has been implicated in a role in the EMT via TLR4/Interleukin 10 (IL10) cascade. The level of secreted protein acidic and cysteine-rich (SPARC) gene, a regulator of EMT, was reported to be 3-4 fold higher in hybrids of BM-derived cell and melanoma.

Analysis of microenvironment microarray assay revealed that fusion hybrids of colon cancer cells and macrophages exhibited a combination of biases, reflecting properties of both parental cells, including fibronectin, collagen XXIII, vitronectin, potentially providing a broader desmoplastic process in different microenvironment. The investigators' preliminary results of differential expression of genes between fusion hybrids of cancer cells and macrophages with non-fused cancer cells show significant elevation of signal pathways involving inflammation, extracellular matrix degradation and mesenchymal phenotypes etc. Besides, prominent increase in signal regulatory protein (SIRP) family members, a cell-cell communicating system, were also found.

Current treatment result of cancer with desmoplasia is unsatisfactory. It is generally believed that desmoplastic stroma provides cancer cells with cytokines/chemokines to suppress immune surveillance and to enhance malignant progression. Recent clinical trials revealed direct targeting desmoplasia using sonic hedgehog inhibitor lead to a more aggressive phenotype with increased regulatory T cells. On the other hand, depleting macrophage or its recruitment from circulation revealed to be effective in reducing pro-fibrotic cytokines/chemokines and CAFs activity; however, with significant normal tissue toxicity.

From previous investigation and our study, fusion hybrids between cancer cells and macrophages appeared to play important role in promoting cancer desmoplasia as well as malignant progression. The investigator proposed to develop an alternative method to ameliorate cancer desmoplasia by focusing on novel targets interfering fusion between cancer cells and macrophages. The potential candidates were revealed by our preliminary microarray study. eg. Signal regulatory protein (SIRP) signal pathway including SIRPa, a macrophage fusion receptor, which was nearly 5 folds differentially expressed in fusion hybrids. Furthermore, the down-stream molecules including DAP12 (DNAX activating protein), a general macrophage fusion regulator, and protein tyrosine phosphatase (PTPN6), protein tyrosine kinase (PTK2B) were increased 8 folds and 4 folds, respectively, in fusion hybrids.

We proposed to target on SIRPa, and other potential candidate molecules with neutralizing antibodies or silencing mRNA to reduce the incidence of fusion phenomenon in cancer with desmoplasia. By reducing the frequency of tumor heterogeneity and the fibrotic phenotype, we would like to improve the therapeutic outcome of cancer with desmoplasia. The combination effect of anti-fusion agents with other anti-fibrosis agents or immunologic therapy will also be explored

ELIGIBILITY:
Inclusion Criteria:

prospective

1. normal peripheral blood laboratory results within one week.
2. hematopoietic cell growth factors are allowed for peripheral blood stem cell donors.
3. hyperemia patients. .
4. age 20 to 70.

retrospective

1. recipient of bone marrow transplantation and developed malignant tumor after transplantation.
2. tumor was resected or biopsied and preserved in Pathology Department. 4-8um thick, 10 slices.

Exclusion Criteria:

prospective

1. malignant cancer patients with no recurrent disease for less than 5 years
2. major cardiovascular disease, immnologic disease, pregnancy.
3. long term users of immuno-suppressants and steroids.

retrospective

(1)none.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: prospectively collect peripheral mononuclear cells: 30 healthy volunteer including peripheral blood stem cell donors, hyperemia.
  Retrospectively collect tumor tissue: 20 patients. malignant cancer patients with history of receiving bone marrow transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
donor derived genes in recipients' tumor tissue | 0-30 years
  Y chromosome and short tandem repeat study of recipients' tumor tissue and donor blood

CONTACTS AND LOCATIONS:
Overall Officials: Ming Yao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Institute of Cancer Research, National Health Research Institutes, Miaoli, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
We will share the data once we publish the results

DOCUMENTS (2):
  • Study Protocol (2022-03-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT05399719/Prot_000.pdf
  • Informed Consent Form (2022-02-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT05399719/ICF_001.pdf